CLINICAL TRIAL: NCT06548373
Title: Assessment of Diagnostic Adequacy of Artificial Intelligence-assisted Point-of-Care Echocardiography Among Anesthesiology Trainees
Brief Title: Assessment of Diagnostic Adequacy of AI-assisted Point-of-Care Echocardiography Among Anesthesiology Trainees
Status: Active, not recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 5240271
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: echocardiography; Artificial Intelligence; AI-assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Year 2 Residents: Loma Linda University Post-Graduate Year 2 Anesthesiology residents providing anesthetic care.
  Interventions: Diagnostic Test: Artificial Intelligence-assisted Point-of-Care Echocardiography

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence-assisted Point-of-Care Echocardiography — A wireless, AI-guided handheld ultrasound probe will be used on adult male patients who present with a clinical indication for peri-anesthesia point-of-care echocardiography examination.
  Residents will document personal interpretation of the completed point-of-care ultrasound (POCUS) examination, important clinical findings, and assessment of whether obtaining a formal echocardiogram is warranted on an exam assessment form. The residents will complete 11 examinations with 10 specific scans each. The first 10 examinations will be AI-guided, and the final 11th examination will be done via a standard (non-AI guided) ultrasound system to gauge the resident's growth in point-of-care echocardiography skill.

SUMMARY:
This pilot study serves to assess the diagnostic adequacy of Artificial Intelligence (AI)-guided point-of-care. Focused echocardiography examinations will be obtained by Anesthesiology trainees and assessed by an expert Cardiologist Echocardiographer. AI-guided echocardiography examinations will be compared to each other. AI-guided and non-AI-guided echocardiography examinations will also be compared.

DETAILED DESCRIPTION:
This pilot study will involve Post-Graduate Year 2 Anesthesiology trainees on rotation in the Loma Linda University Medical Center operating rooms. Prior to participation, the trainees will give written informed consent to participate in the study and complete a baseline questionnaire to collect information regarding prior education in point-of-care echocardiography and the number of those examinations personally performed prior to study participation. All subjects will watch a brief training video about the AI guidance platform and participate in a hands on training session to familiarize themselves with AI guidance.

When adult patients having anesthesia for procedures present with a clinical indication for peri-anesthesia point-of-care echocardiography examination, the assigned trainee will use the AI-guided system to obtain a standardized point-of-care focused cardiac examination. Subjects will be completing 11 total examinations, 10 using AI guidance, 1 without.

Images of the examination will be assessed by an expert Cardiologist Echocardiographer that is blinded to the resident involved to measure diagnostic adequacy.

A final non-AI-guided echocardiogram examination will be completed by the resident to measure and compare the time and adequacy of the images to the AI-guided examination images.

ELIGIBILITY:
Inclusion Criteria:

* Loma Linda University resident in Anesthesiology
* Post-Graduate Year 2

Exclusion Criteria:

* Residents not a part of a Loma Linda University residency program
* Residents not a part of an Anesthesiology residency program
* Loma Linda University Anesthesiology Post-Graduate Year 1 Residents
* Loma Linda University Anesthesiology Post-Graduate Year 3 Residents
* Loma Linda University Anesthesiology Post-Graduate Year 4 Residents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes Loma Linda University 2024 - 2025 Post-Graduate Year 2 Anesthesiology residents providing anesthetic care.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Echocardiogram Evaluation | Within 24 hours of AI-guided examination completion
  Cardiologist will review AI-assisted echocardiogram images obtained by residents for diagnostic image quality. A rating of "Yes" will represent a diagnostically accurate result and a rating of "No" will represent an image that is not adequate for diagnostic purposes.

SECONDARY OUTCOMES:
Change in length of time of AI-assisted echocardiogram procedure | Change in time of individual examination completion between the first AI-guided echocardiography examination performed and the tenth AI-guided echocardiography examination performed, typically one month post-enrollment
  Assessment of time to complete the standardized point-of-care focused echocardiography examination will be determined by comparing time stamps on the first and last image sequence recorded. Change in this interval will be assessed between the tenth and first studies performed.
Change in echocardiogram examination image quality through comparison of AI-guided and non-AI-guided echocardiogram examination | Change in time between the tenth AI-guided echocardiography examination performed and the non-AI guided cardiography examination performed, typically two months post-enrollment
  After the 10th AI-guided point-of-care focused echocardiography examination is completed, the trainee will complete a standardized point-of-care focused echocardiography examination using a standard (not AI-guided) system. Assessment of echocardiogram adequacy, time to complete the examination, and Concordance between the trainee and Cardiologist assessments will be analyzed as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate, MD, Study Chair — Loma Linda University
Locations (1):
- Loma Linda University Troesch Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofer CK, Mizuguchi AK, Popescu WM. Monitoring the patient at risk of hemodynamic instability in remote locations. Int Anesthesiol Clin. 2012 Spring;50(2):141-72. doi: 10.1097/AIA.0b013e318250ebb1. No abstract available. PMID 22481561
- [Background] Kratz T, Steinfeldt T, Exner M, Dell Orto MC, Timmesfeld N, Kratz C, Skrodzki M, Wulf H, Zoremba M. Impact of Focused Intraoperative Transthoracic Echocardiography by Anesthesiologists on Management in Hemodynamically Unstable High-Risk Noncardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):602-609. doi: 10.1053/j.jvca.2016.11.002. Epub 2016 Nov 2. PMID 28089598
- [Background] Staudt GE, Shelton K. Development of a Rescue Echocardiography Protocol for Noncardiac Surgery Patients. Anesth Analg. 2019 Aug;129(2):e37-e40. doi: 10.1213/ANE.0000000000003569. PMID 29916865
- [Background] Via G, Hussain A, Wells M, Reardon R, ElBarbary M, Noble VE, Tsung JW, Neskovic AN, Price S, Oren-Grinberg A, Liteplo A, Cordioli R, Naqvi N, Rola P, Poelaert J, Gulic TG, Sloth E, Labovitz A, Kimura B, Breitkreutz R, Masani N, Bowra J, Talmor D, Guarracino F, Goudie A, Xiaoting W, Chawla R, Galderisi M, Blaivas M, Petrovic T, Storti E, Neri L, Melniker L; International Liaison Committee on Focused Cardiac UltraSound (ILC-FoCUS); International Conference on Focused Cardiac UltraSound (IC-FoCUS). International evidence-based recommendations for focused cardiac ultrasound. J Am Soc Echocardiogr. 2014 Jul;27(7):683.e1-683.e33. doi: 10.1016/j.echo.2014.05.001. PMID 24951446
- [Background] Shillcutt SK, Markin NW, Montzingo CR, Brakke TR. Use of rapid "rescue" perioperative echocardiography to improve outcomes after hemodynamic instability in noncardiac surgical patients. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):362-70. doi: 10.1053/j.jvca.2011.09.029. Epub 2012 Jan 4. PMID 22226417